CLINICAL TRIAL: NCT06862986
Title: The Effect of Ear Massage on Bowel Activity in Patients Undergoing Lower Extremity Surgery: A Randomized Controlled Study
Brief Title: Ear Massage Effect on Bowel Activity After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, sumbule koksoy vayisoglu, PhD , Department of Public Health Nursing, Principal investigator, Assoc. Prof. Dr., Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EarMassageMersinU
Record Dates: First submitted 2025-03-05; First posted 2025-03-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Constipation; Lower Extremity Surgery
Keywords: Ear massage; lower extremity surgery; constipation; bowel activity
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, Two-arm, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the clinic where the study was conducted, patients who will undergo lower extremity surgery are placed on bed rest and restricted movement before surgical intervention and hospitalized in the clinic for approximately one day to ensure optimum preparation of the patient for surgery. During this period, the constipation status of the patients before surgical intervention is evaluated and if the patients state that they are unable to defecate, an enema is administered to ensure defecation before surgical intervention. After surgical intervention, patients are on absolute bed rest for 24 hours and their first mobilization is provided upon physician's request. In this period, the first gas and defecation time of the patients are routinely recorded by the nurses in the ward, and enemas (sodium phosphate) and laxatives (lactulose) are administered to patients who do not have gas and defecation in the first 3 days after surgical intervention. In the study, no procedure other than routine t
- Ear massage group (Experimental): At least one Intervention must be specified for an Interventional study. Patients included in the study group will receive ear massage in addition to the routine treatment and care practices of the clinic. Ear massage application will be started in the evening of the first day after surgical intervention (at 19:30) and will be applied twice a day at least 30 minutes after morning and evening meals (07:30 am, 19:30 pm) for 3 minutes each, similar to the literature (8,9,12). The bowel sounds of the patients will be re-evaluated before and 10 minutes after the ear massage application, and the excretory activities form will be filled out. Ear massage application will be terminated when the patient defecates or when the patient is given an enema.
  Interventions: Other: Ear massage

INTERVENTIONS:
Other: Ear massage — At least one Intervention must be specified for an Interventional study. Patients included in the study group will receive ear massage in addition to the routine treatment and care practices of the clinic. Ear massage application will be started in the evening of the first day after surgical intervention (at 19:30) and will be applied twice a day at least 30 minutes after morning and evening meals (07:30 am, 19:30 pm) for 3 minutes each, similar to the literature (8,9,12). The bowel sounds of the patients will be re-evaluated before and 10 minutes after the ear massage application, and the excretory activities form will be filled out. Ear massage application will be terminated when the patient defecates or when the patient is given an enema.
  Arms: Ear massage group

SUMMARY:
Constipation is seen in patients undergoing orthopedic surgical interventions at rates as high as 23% to 94%. Constipation develops more frequently in individuals undergoing major orthopedic surgical interventions such as lower extremity arthroplasties and lower extremity fracture repairs. Ear massage is one of the methods that is thought to be effective in preventing or reducing constipation that may develop in the early period by activating the parasympathetic nervous system after surgical intervention, increasing intestinal peristalsis and emptying the intestinal contents. The ear both contains its own unique points and is directly or indirectly connected to 12 body meridians. Massage applied to the ear provides balance between vital energy (qi) and blood flow (yin-yang) (12). The qi of the person stimulated by massaging these points in the ear is connected to certain organs such as the intestines through channels or meridians. Thanks to this connection, bowel movements can be stimulated and constipation can be eliminated. Ear massage has the potential to be an effective non-pharmacological method for the relief of gastrointestinal problems such as constipation.

DETAILED DESCRIPTION:
Constipation, which frequently develops after surgical intervention and is an undesirable problem, is seen at high rates ranging from 23% to 94% in patients undergoing orthopedic surgical intervention. This rate varies according to the type of surgical intervention performed and is higher especially in individuals undergoing major orthopedic surgical interventions such as lower extremity arthroplasties and lower extremity fracture repairs. Patients undergoing lower extremity surgery have mobility limitations before and after surgical intervention, prolonged fasting before surgical intervention, dietary changes, surgical intervention performed under general anesthesia, opioid/nonopioid analgesia used in pain management, inability to take the appropriate position for defecation, use of bedpan, and applications such as plaster, traction, joint prosthesis that cause limitation of movement cause constipation in patients. Constipation causes patients to face many physiologic and psychologic problems such as restlessness, abdominal tension, epigastric pain, diaphragmatic tension, hypotension, tachycardia and delays postoperative recovery.

Ear massage is one of the methods that is thought to be effective in preventing or reducing constipation that may develop in the early period by activating the parasympathetic nervous system, increasing intestinal peristalsis and emptying the intestinal contents after surgical intervention. Anatomically, the ear is an organ with dense vessels and nerves and the only peripheral branch of the vagus nerve is located in the outer ear. Stimulation of the points on the vagus nerve in the ear with ear massage can directly activate the parasympathetic nervous system. With the activation of the parasympathetic nervous system, the neural networks in the digestive system, especially the vagovagal neurocircuits, become more active. With the activation of vagovagal neurocircuits, the enteric nervous system (ENS), which provides independent functioning of the intestines and other gastrointestinal organs, is activated. The ENS, whose activation increases with this interaction, regulates electrical and chemical transmission in the digestive tract and helps the intestines to function more efficiently.

On the other hand, the ear is one of the most important organs in Traditional Chinese Medicine. The ear both contains its own specific points and is directly or indirectly connected to 12 body meridians. Massage applied to the ear ensures balance between vital energy (qi) and blood flow (yin-yang). The qi of the person stimulated by massaging these points in the ear is connected through channels or meridians to specific organs such as the intestines. This connection stimulates bowel movements and relieves constipation.

Ear massage has the potential to be an effective non-pharmacologic method for the relief of gastrointestinal problems such as constipation. Although there are studies in the literature showing that massages applied to different areas such as the abdomen in patients undergoing orthopedic surgery have a positive effect on gastrointestinal system functions, there is no study examining the effect of ear massage on the excretory activities of patients undergoing lower extremity surgery. Based on the aforementioned information, the aim of this study was to determine the effect of ear massage on excretory activities (return time of bowel sounds, time to first defecation, number of bowel sounds and number of laxative use) in patients undergoing lower extremity surgery, who were at high risk for the development of constipation after surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Not signing the Informed Volunteer Consent Form,
* Under 18 years of age and over 65 years of age,
* Unconscious or having problems with orientation,
* Those who cannot speak Turkish and do not understand it,
* undergoing surgical intervention at sites other than the lower extremities,
* Physician-diagnosed chronic constipation or history of diseases that may affect intestinal peristalsis (inflammatory bowel disease, presence of abdominal tumor, surgical intervention or radiotherapy to the abdominal region, presence or suspicion of ileus, and pregnancy) and regular laxative users,
* Enemas administered before surgical intervention,
* Patients who have problems with the transition to oral feeding and who are unable to feed orally will be included in the study.

Exclusion Criteria:

* Not signing the Informed Volunteer Consent Form,
* Under 18 years of age and over 65 years of age,
* Unconscious or having problems with orientation,
* Those who cannot speak Turkish and do not understand it,
* undergoing surgical intervention at sites other than the lower extremities,
* Physician-diagnosed chronic constipation or history of diseases that may affect intestinal peristalsis (inflammatory bowel disease, presence of abdominal tumor, surgical intervention or radiotherapy to the abdominal region, presence or suspicion of ileus, and pregnancy) and regular laxative users,
* Enema administered before surgical intervention,
* Patients who have problems with transition to oral feeding and who cannot be fed orally will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Time for the return of the bowel sound | Up to three days
  The time of the first return of the bowel sounds of the patients after the surgical intervention will be recorded by asking the researcher by asking twice a day (morning-evening).
First defecation time after surgery | Up to three days
  The time of the patients' first defecation time after surgical intervention will be recorded by asking the investigator by asking twice a day (morning-evening).

SECONDARY OUTCOMES:
the number of bowel sounds | up to three days
  After the surgical intervention, the number of bowel sounds of the patients will be recorded twice a day (morning and evening) by the investigator.
use of defecation aids | up to three days
  After the surgical intervention, the patients' use of defecation aids will be recorded by the investigator by asking them twice a day (morning-evening).

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to avoid duplication, it is not intended to be shared until the research is completed.

REFERENCES:
- [Result] Yue C, Liu Y, Zhang X, Xu B, Sheng H. Randomised controlled trial of a comprehensive protocol for preventing constipation following total hip arthroplasty. J Clin Nurs. 2020 Aug;29(15-16):2863-2871. doi: 10.1111/jocn.15299. Epub 2020 May 26. PMID 32320100
- [Result] Jiang ZF, Liu G, Sun XX, Zhi N, Li XM, Sun R, Zhang H. Auricular acupressure for constipation in adults: a systematic review and meta-analysis. Front Physiol. 2023 Oct 16;14:1257660. doi: 10.3389/fphys.2023.1257660. eCollection 2023. PMID 37908337
- [Result] Kuo SY, Tsai SH, Chen SL, Tzeng YL. Auricular acupressure relieves anxiety and fatigue, and reduces cortisol levels in post-caesarean section women: A single-blind, randomised controlled study. Int J Nurs Stud. 2016 Jan;53:17-26. doi: 10.1016/j.ijnurstu.2015.10.006. Epub 2015 Oct 22. PMID 26525188
- [Result] Tseng YT, Chen IH, Lee PH, Lin PC. Effects of auricular acupressure on depression and anxiety in older adult residents of long-term care institutions: A randomized clinical trial. Geriatr Nurs. 2021 Jan-Feb;42(1):205-212. doi: 10.1016/j.gerinurse.2020.08.003. Epub 2020 Sep 11. PMID 32921508
- [Result] Jing X, Liu J, Wang C, Ji M, Chen X, Mei Y, Zhu QR. Auricular acupressure is an alternative in treating constipation in leukemia patients undergoing chemotherapy: A systematic review and meta-analysis. Complement Ther Clin Pract. 2018 May;31:282-289. doi: 10.1016/j.ctcp.2018.03.005. Epub 2018 Mar 14. PMID 29705469
- [Result] Nouhi E, Mansour-Ghanaei R, Hojati SA, Chaboki BG. The effect of abdominal massage on the severity of constipation in elderly patients hospitalized with fractures: A randomized clinical trial. Int J Orthop Trauma Nurs. 2022 Nov;47:100936. doi: 10.1016/j.ijotn.2022.100936. Epub 2022 Feb 24. PMID 36274468
- [Result] Seyyedrassoli, A., Ghahramanian, A., Azizi, A., Goljarian, S., Gillespie, M., & Aydinferd, S. (2018). Comparison of effectiveness of reflexology and abdominal massage on constipation among orthopedic patients: A single-blind randomized controlled trial. International Journal of Medical Research & Health Sciences, 5
- [Result] Lee TH, Lee JS, Hong SJ, Jang JY, Jeon SR, Byun DW, Park WY, Kim SI, Choi HS, Lee JC, Lee JS. Risk factors for postoperative ileus following orthopedic surgery: the role of chronic constipation. J Neurogastroenterol Motil. 2015 Jan 1;21(1):121-5. doi: 10.5056/jnm14077. PMID 25537675
- [Result] G Rler H, Y Ld Z FT, Bekmez F. A Common Complication in Orthopedic Patients: Postoperative Constipation and Related Risk Factors. J Perianesth Nurs. 2023 Oct;38(5):e15-e20. doi: 10.1016/j.jopan.2023.05.004. Epub 2023 Aug 12. PMID 37578408